CLINICAL TRIAL: NCT02960789
Title: Hydration Status Evaluation on Admittance and During Rehydration of Dehydrated Children at Boston Children's Hospital, With Exploratory Hydration Assessment Devices
Brief Title: Hydration Status Evaluation of Dehydrated Children With Experimental Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Boston Children's Hospital (Other); National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 1606619184; U54EB015408 (NIH)
Record Dates: First submitted 2016-11-04; First posted 2016-11-10 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2018-12

CONDITIONS: Dehydration
Keywords: Dehydration; Children; Measurement
MeSH Terms: conditions — Dehydration

ARMS (1):
- Dehydrated Children (Experimental): Children between the ages of 2 to 18 years of age presenting to the Emergency Department at Children's Hospital Boston with complaints such as "Dehydration", "Gastroenteritis", "Vomiting", and or "Intolerance of POs" be approached by study personnel for possible participation in the study.
  Interventions:
  * Undertake and record a formalized clinical assessment of hydration status
  * Take a measurement of body weight on calibrated scales
  * "RF wristband" hydration status measurement
  * Measure capillary refill time with manual stopwatch
  * "CRT device" hydration status measurement
  Interventions: Other: Formalized clinical assessment of hydration status; Other: Take a measurement of body weight on calibrated scales; Device: "RF wristband" hydration status measurement; Other: Measure capillary refill time with manual stopwatch; Device: "CRT device" hydration status measurement

INTERVENTIONS:
Other: Formalized clinical assessment of hydration status — Undertake and record a standard formalized clinical hydration assessment
Other: Take a measurement of body weight on calibrated scales — Standard body weight measurements conducted on calibrated scales
Device: "RF wristband" hydration status measurement — Take measurements with "RF wristband" radio-frequency non-invasive wrist-based hydration status assessment device
Other: Measure capillary refill time with manual stopwatch — A standard visual assessment of capillary refill time, aided by the use of a stopwatch
Device: "CRT device" hydration status measurement — Take measurements with "CRT device" for non-invasively quantitatively assessing Capillary Refill Time

SUMMARY:
A pediatric study in collaboration with Boston Children's Hospital to review the performance of two novel hydration status measurement devices against standard clinical assessment methods, through repeated measurement of hydration status of dehydrated children admitted to the emergency department receiving rehydration therapy, followed by an at-home follow-up measurement once symptoms have resolved.

DETAILED DESCRIPTION:
This is a prospective cohort study to determine the performance of two prototype devices developed to aid in the diagnosis and monitoring of physiological hydration state of dehydrated children. These children are patients presenting to the emergency department with varying degrees of dehydration.

Overview of study procedure:

1. Initial identification of eligible patients. Patients will be initially identified by their chief complaint after registration and triage. Terms such as "Dehydration", "Gastroenteritis", "Diarrhea", "Vomiting", and or "Intolerance of POs" will be noted and those patients will be approached by study personnel for possible participation in the study.
2. Screening and obtaining of consent After patients have been identified as meeting entry criteria for the study, the parents will be asked two screening questions: 1. How far of a distance do you live from the hospital? 2. Would you be interested in a study that includes a follow-up home visit? These questions will be used to gauge the ability of the family to realistically complete the study, as a research coordinator will be travelling to the home to conduct a follow up visit after symptom resolution.
3. Study enrollment i. Risks and benefits of study participation will be discussed, as well as the consent process. After consent is obtained, a symptom survey will be administered to each patient and family to determine the degree of dehydration based on clinical assessment. Detailed information regarding onset and degree of symptoms including vomiting, diarrhea, urine output and amount of oral fluid intake will be recorded. A similar survey was administered as part of a randomized control trial of Dextrose containing fluids, which was conducted in our Emergency Department, (Levy, Waltzman).

   ii. Each patient will have his/her weight obtained using a calibrated digital scale in a dry diaper or underwear with an appropriately sized gown. Then both study devices will be utilized by study personnel to obtain three triplicate measurements. Replicate measurements of capillary refill times will also be obtained in the same locations by visual inspection using a commercial stopwatch. Additional information including ambient room temperature, patient skin temperature and amount of applied pressure during the Capillary Refill Time measurements will be recorded.

   iii. After the initial measurements are obtained, the treating provider will be given a questionnaire outlining their assessment of the degree of dehydration of the patient and the study protocol. Patients will be treated per the discretion of the health care provider including admission to the hospital or discharge based on his or her clinical judgment. Device measurements will not be provided to the treating clinician. Measurements obtained from the device will have no bearing on the clinical treatment of the patients. All measurements obtained in relation to the study will be used solely for research purposes. Device measurements of capillary refill time and radio-frequency measurements, and initial weight will not be disclosed to treating staff.

   iv. Prior to either discharge from the emergency department or admission to the hospital, each participating family will be given a symptom log to serve as a method for objectively tracking degree of symptoms during the follow up period.
4. Initial follow up and monitoring of symptom resolution:

   A research coordinator will call each patient's family by phone within 24-72 hours after initial enrollment. He or she will establish contact with the family and explain the follow up plan and monitoring for symptom resolution. Regular follow up by phone every 48 hours will continue until the symptoms have resolved; at which time an in-person follow up visit will be planned within 24-72 hours.
5. In-person follow-up After the resolution of symptoms (vomiting and/or diarrhea), the research coordinator will travel to the residence of each patient and repeat the measurements including weight and device measurements. Again the weight will be performed on a calibrated digital scale with the patient in a dry diaper or underwear and an appropriately sized gown. Also, the study coordinator will ask the family/patient to answer questions related to the duration of the illness, and other visits with medical providers that have occurred in the interim. The radio-frequency and capillary refill time measurements will be stored in a secure de-identified server, and all remaining data will be recorded entered into a password-protected digital database using RedCap.

ELIGIBILITY:
Inclusion Criteria:

Dehydrated children, indicated primarily by chief complaints or symptoms of vomiting, diarrhea, dehydration, gastroenteritis or intolerance of oral intake for less than or equal to 5 days

Exclusion Criteria:

1. Previously enrolled in this study
2. Children with a pre-existing medical condition which may potentially affect either the course or nature of their current illness, or a skin condition which has the potential to alter their capillary refill time, specifically:

   a. Pre-existing medical conditions i. Immunosuppression (HIV, malignancy) ii. Existing gastrointestinal condition (Inflammatory bowel disease, Crohns disease, ulcerative colitis, or recent abdominal surgery within prior 30 days) iii. Uncorrected or palliated cardiac disease iv. Other chronic medical condition other than asthma or eczema (such as cystic fibrosis, diabetes, or patients with an indwelling devices such as gastrostomy, nasogastric or nasojejunal tube, or ventriculoperitoneal shunts

   b. Concern for surgical abdomen i. Abdominal trauma or head trauma as reason for visit ii. Potential surgical condition (concern for appendicitis, intussusception, malrotation, volvulus, bowel obstruction)

   c. Skin condition which may alter optical and radio-frequency measurements, or cause discomfort i. Acanthosis ii. Severe eczema covering all exposed testing sites to measure capillary refill iii. Burns

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2016-11; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight (Weight at follow-up visit minus weight in emergency department) | 1-14 days
Change in capillary refill time as measured by experimental measurement device 1. | 1-14 days
Change in wrist water content as measured by experimental measurement device 2. | 1-14 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts